CLINICAL TRIAL: NCT02464306
Title: Fidaxomicin Versus Standard of Care Therapy in Solid Organ Transplant Recipients With Clostridium Difficile Infection
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lost funding
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-2257
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Clostridium Difficile Infection; Solid Organ Transplant
Keywords: recipients
MeSH Terms: conditions — Clostridium Infections | interventions — Fidaxomicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SOT Recipients (Experimental): SOT recipients (heart, lung, kidney, liver, kidney-pancreas, and pancreas) with a first-episode of CDI. Patients will be treated with fidaxomicin 200 mg PO twice daily for 10 days. The rate of sustained clinical response (SCR; cure without recurrence at 30 days) will be assessed.
  Interventions: Drug: fidaxomicin
- Historical Cohort (No Intervention): Historical cohort of SOT recipients who received standard of care therapy for CDI at our institution.

INTERVENTIONS:
Drug: fidaxomicin — Patients will be treated with fidaxomicin 200 mg PO twice daily for 10 days.
  Arms: SOT Recipients

SUMMARY:
A prospective study to assess the efficacy and safety of fidaxomicin in Solid Organ Transplant (SOT) recipients (heart, lung, kidney, liver, kidney-pancreas, and pancreas) with a first-episode of Clostridium difficile infection (CDI).

DETAILED DESCRIPTION:
Patients will be treated with fidaxomicin 200 mg PO twice daily for 10 days. The rate of sustained clinical response (SCR; cure without recurrence at 30 days) will be assessed and compared to a historical cohort of SOT recipients who received standard of care therapy for CDI at our institution. The data for the historical control group will be collected under a separate IRB-approved protocol. Standard of care therapy will be considered oral or intravenous metronidazole and / or oral vancomycin. The study will be powered to show non-inferiority of fidaxomicin compared to standard of care treatment in SOT recipients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater and up 85 years
* SOT recipient (lung, heart, kidney, liver, kidney-pancreas, pancreas)
* First episode of CDI

Exclusion Criteria:

* Receiving additional therapies with activity again C. difficile (oral bacitracin, fusidic acid, and/or rifaximin)
* Toxic megacolon
* Ileus or significant abdominal distension
* Hypotension with vasopressor requirement
* History of inflammatory bowel disease
* Pregnancy
* Decisionally challenged
* Prisoners
* >4 doses of metronidazole for the treatment of C. difficile in the previous 7 days
* >4 doses of oral vancomycin in the previous 7 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a sustained clinical response (SCR), defined as clinical cure with no recurrence. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Kelly E Schoeppler, PharmD, Principal Investigator — University of Colorado, Denver